CLINICAL TRIAL: NCT02284971
Title: A Pilot Study to Assess the Combination of Stereotactic Body Radiation Therapy and CDX-1127 in Modulating Local and Systemic T-cell Responses Against Prostate Cancer
Brief Title: Pilot Study of SBRT and CDX-1127 in Prostate Cancer
Acronym: Prostate-04
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accruals
Sponsor: James Larner, MD (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, James Larner, MD, Professor, Radiation Oncology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17456
Record Dates: First submitted 2014-10-29; First posted 2014-11-06 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — varlilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: CDX1127 & SBRT Concurrent (Experimental): SBRT will be administered to the primary tumor and/or site of metastatic disease over a period of 5 days (Days 1-5) at a constant dose for 1-4 sites of prostate cancer involvement:30 Gy in 5 fractions of 6 Gy each for prostate gland; 25 Gy in 5 fractions for bone and/or soft tissue metastases).
  Subjects will receive four doses of CDX-1127(3 mg/kg) (Days 1, 43, 64, 85). The study drug will be administered intravenously over a 90-minute time period and will be followed by a 2-hour observation period. A subject's dose of CDX-1127 will be calculated based on their actual body weight at the time of screening. A subject's dose of CDX-1127 will remain constant at each time point, unless they experience a greater than 10% change in body weight.
  Interventions: Biological: CDX1127; Radiation: SBRT
- Arm B: CDX1127 & SBRT Sequential; CDX1127 upfront (Experimental): SBRT will be administered to the primary tumor and/or sites of metastatic disease over a period of 5 days (Days 22-26) at a constant dose for 1-4 sites of prostate cancer involvement:30 Gy in 5 fractions of 6 Gy each for prostate gland; 25 Gy in 5 fractions for bone and/or soft tissue metastases).
  Subjects will receive four doses of CDX-1127(3 mg/kg) (Days 1, 43, 64, 85). The study drug will be administered intravenously over a 90-minute time period and will be followed by a 2-hour observation period. A subject's dose of CDX-1127 will be calculated based on their actual body weight at the time of screening. A subject's dose of CDX-1127 will remain constant at each time point, unless they experience a greater than 10% change in body weight.
  Interventions: Biological: CDX1127; Radiation: SBRT
- Arm C: CDX1127 & SBRT Sequential; SBRT upfront (Experimental): SBRT will be administered to the primary tumor and/or sites of metastatic disease over a period of 5 days (Days 1-5) at a constant dose for 1-4 sites of prostate cancer involvement:30 Gy in 5 fractions of 6 Gy each for prostate gland; 25 Gy in 5 fractions for bone and/or soft tissue metastases).
  Subjects will receive four doses of CDX-1127(3 mg/kg) (Days 22, 43, 64, 85). The study drug will be administered intravenously over a 90-minute time period and will be followed by a 2-hour observation period. A subject's dose of CDX-1127 will be calculated based on their actual body weight at the time of screening. A subject's dose of CDX-1127 will remain constant at each time point, unless they experience a greater than 10% change in body weight.
  Interventions: Biological: CDX1127; Radiation: SBRT

INTERVENTIONS:
Biological: CDX1127
  Other Names: Varlilumab
Radiation: SBRT

SUMMARY:
This study evaluates the combination of stereotactic body radiation therapy (SBRT) and CDX-1127 in subjects with castration resistant prostate cancer. Subjects will be randomized to one of three arms to receive SBRT prior to, after, or in conjunction with the first dose of CDX-1127.

DETAILED DESCRIPTION:
This pilot study will be conducted in subjects with metastatic prostate cancer in order to define whether inclusion of immune regulation agents such as CDX-1127 augments immune responses to SBRT-treated primary tumors or metastases, and whether inclusion of CDX-1127 in the treatment regimen results in immune responses in untreated metastases.

ELIGIBILITY:
MAIN INCLUSION CRITERIA

Males, Age ≥ 18 years.

Participants must have histologically-proven prostrate adenocarcinoma that is castrate-resistant. Progressive disease is defined by one or more of the following:

* A rise in PSA on two successive determinations at least one week apart and PSA level ≥2ng/ml.
* Soft-tissue progression defined by RECIST 1.1.
* Bone disease progression defined by PCWG2 with two or more new lesions on bone scan.

Patients must have castrate levels of testosterone (<50 ng/dl [1.74 nmol/l]).

Patients must have undergone orchiectomy, or have been on LHRH agonists or antagonists, for at least 3 months prior to drug initiation. Patients on LHRH agonists/antagonists must remain on these agents for the duration of the study.

Clinical metastases must be present and confirmed on imaging studies.

Participants for whom radiation therapy is recommended for the prostate gland (or prostate bed nodule) and/or bone or soft tissue metastases.

SBRT may be administered to 1-4 sites and the treatment sites can include prostate gland (or prostate bed nodule for post-prostatectomy patients), bone metastases, and soft tissue metastases. Participants must have at least one site of disease that will be both irradiated with SBRT and biopsied to evaluate immunological outcomes.

ECOG performance status 0-2.

Adequate hepatic and renal function.

MAIN EXCLUSION CRITERIA

Prior malignancies, that will affect the completion and interpretation of the study.

Patients with active CNS metastases from prostate cancer.

Patients who are currently receiving systemic cytotoxic chemotherapy, radiation, or other experimental therapy, or who have received this therapy within the preceding 4 weeks. Patients who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks are excluded.

Patients who are currently receiving systemic cytotoxic chemotherapy, radiation, or other experimental therapy, or who have received this therapy within the preceding 4 weeks.

Major surgery within 4 weeks prior to the start of study treatment.

Patients who are receiving or have previously been treated CDX-1127.

HIV positivity

Evidence of active Hepatitis B virus or Hepatitis C virus.

Patients receiving the following medications at study entry or within the preceding 4 weeks (or longer, if otherwise specified) are excluded:

1. Checkpoint inhibitors (within the preceding12 weeks)
2. Allergy desensitization injections
3. Systemic corticosteroids of more than 10 mg per day of prednisone (or equivalent), administered parenterally or orally, except for physiologic replacement. Inhaled steroids (e.g. Advair®, Flovent®, Azmacort®) are not permitted. Topical corticosteroids are acceptable, including steroids with very low solubility administered nasally for local effects only (e.g. Nasonex®)
4. Any growth factors (e.g. GM-CSF, G-CSF, erythropoietin).
5. Interferon or interleukin therapy
6. Other Agents with putative immunomodulating activity. (e.g. sipuleucel-T (Provenge ®))

Other investigational drugs or investigational therapy if the patient is currently taking those drugs/therapy, or if they have received the drugs/therapy within 4 weeks prior to the start of study treatment.

Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement.

Significant cardiovascular disease.

Active bleeding disorders or evidence of chronic or acute disseminated intravascular coagulation (DIC).

Concomitant therapeutic anticoagulation (i.e., warfarin) for reasons other than venous catheter patency.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to day 270
Immunologic (CD8+ T cell and T regulatory cell (Treg) infiltration) | Up to day 43
  • Estimate the effect of SBRT, CDX-1127 and the combination of SBRT and CDX- 1127 on CD8+ T cell and T regulatory cell (Treg) infiltration in prostate tumors.

SECONDARY OUTCOMES:
Immunologic (lymphocyte composition of blood over time). | Up to day 270
  • Estimate the effect of SBRT, CDX-1127, and the combination of SBRT and CDX-1127 on the lymphocyte composition of blood over time.

CONTACTS AND LOCATIONS:
Overall Officials: James Larner, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States